CLINICAL TRIAL: NCT03794700
Title: Pilot Evaluation of Hospice Decision Support Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-1138; 1R21AG059114-01 (NIH)
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hospice; End-of-life Decision Making; Hospice Decision Making
Keywords: Hospice; End-of-life; Patient decision aid; Shared decision making
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Other): Participants will receive hospice decisional support materials and be asked to review them. Participants will provide feedback on tools and complete feasibility, efficacy and knowledge assessments.
  Interventions: Other: Hospice Decision Aids

INTERVENTIONS:
Other: Hospice Decision Aids — Paper and video hospice decision aid
  Arms: Intervention

SUMMARY:
The goal of this project is to determine the feasibility and acceptability of a hospice decision aid among a diverse population of older adults at multiple stages of illness (Aim 1) and to determine the preliminary efficacy of the hospice decision aid on decision quality, hospice knowledge, and values-concordance (Aim 2). By testing the feasibility, acceptability, and preliminary efficacy of a novel hospice Patient Decision Aid (PTDa) in a diverse population of older adults, additionally the study will simultaneously explore barriers to PtDA implementation in both an outpatient primary care and inpatient palliative care setting. The study will also gather sufficient pilot data to support a subsequent effectiveness/implementation trial and thus address the absence of quality of SDM interventions for end-of-life care decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 65 or older.
* At least one life-limiting illness or syndrome.

Exclusion Criteria:

* Non-English speakers.
* Patients with cognitive Impairments preventing ability to provide informed consent.
* Patients on isolation precautions due to resistant bacteria or impaired immune function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Matlock, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brereton E, Harger G, Matlock DD, Dorsey Holliman B, Tate CE. How Do Patients Describe Hospice Care? A Qualitative Analysis of the Language Used by Older Adults to Describe Hospice Care. J Palliat Med. 2022 Nov;25(11):1692-1696. doi: 10.1089/jpm.2022.0011. Epub 2022 Aug 9. PMID 35944273
- [Derived] Tate CE, Venechuk G, Pierce K, Khazanie P, Ingle MP, Morris MA, Allen LA, Matlock DD. Development of a Decision Aid for Patients and Families Considering Hospice. J Palliat Med. 2021 Apr;24(4):505-513. doi: 10.1089/jpm.2020.0250. Epub 2021 Jan 13. PMID 33439075

RESULTS

PARTICIPANT FLOW:
Groups:
- No Hospice Decision Aid: Did not receive the intervention (i.e. Hospice Decision Aid)
- Hospice Decision Aid: Participants will receive hospice decisional support materials and be asked to review them. Participants will provide feedback on tools and complete feasibility, efficacy and knowledge assessments.
  Hospice Decision Aids: Paper and video hospice decision aid
Period: Overall Study
Arm/Group | No Hospice Decision Aid | Hospice Decision Aid
Started | 43 | 88
Completed | 43 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants did not review the intervention (i.e. Hospice Decision Aid)
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 43 | 88 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 43 | 88 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 56 | 84
  Male | 15 | 32 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 28 | 69 | 97
  Unknown or Not Reported | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 43 | 88 | 131
Hospice Knowledge Test [Mean (Full Range); unit: units on a scale] — Hospice knowledge was quantitatively assessed using the 23-item hospice knowledge survey.This survey consists of true/false questions, with scores ranging from 0 to 23, awarding one point for each correct answer. A higher score indicates more knowledge of hospice. The Cronbach's α = 0.75 indicates a good degree of internal reliability. Absolute values measured at baseline and one month
  units on a scale | 18 [12 to 23] | 18 [0 to 23] | 18 [0 to 23]
Hospice Beliefs and Attitudes Scale [Mean (Full Range); unit: units on a scale] — The HBAS is an 8-item scale designed to measure beliefs and attitudes regarding hospice care. T Cronbach's α = .74 for the scale, indicating a good degree of internal reliability.The HBAS is scored from 8 to 40, with a higher score indicating more positive views of hospice care. The scale uses a 5-item Likert scale with answers ranging from "strongly disagree" to "strongly agree" for all questions. Absolute values measured at baseline and one month
  units on a scale | 29 [18 to 40] | 29 [12 to 40] | 29 [12 to 40]
Decision Self Efficacy Scale [Mean (Full Range); unit: units on a scale] | 92 [66 to 100] | 87 [0 to 100] | 89 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Hospice Knowledge Scale
Description: Hospice Knowledge Scale is a 23-item true/false scale that measures patient knowledge about hospice care. Each question is worth 1 point with possible scores ranging from 0 to 23. Higher scores indicate more knowledge.
Time Frame: 1 month follow-up
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Control: Did not receive intervention (i.e. Patient Decision Aid)
Arm/Group | Control | Intervention
Number analyzed (Participants) | 43 | 88
score on a scale | 18 [0 to 23] | 17 [0 to 23]

2. Primary Outcome: Hospice Beliefs and Attitudes Scale
Description: 8-item scale developed to measure beliefs and attitudes towards hospice care. It has a Cronbach's α = .74 for the scale, indicating a good degree of internal reliability. Scores from 8 to 40. Higher scores indicate better opinions of hospice. .
Time Frame: 1-Month follow up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 43 | 88
units on a scale | 32 [26 to 40] | 33 [11 to 40]

3. Primary Outcome: Decision Self Efficacy Scale
Description: Is an 11-item instrument that one's self-confidence in decision making. This scale is a validated scale with a Cronbach's alpha of 0.92 and correlates with DCS subscale of being informed (r=0.47). Scored from 0-100 with higher scores indicating more decision self efficacy.
Time Frame: 1 month Follow up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 43 | 88
units on a scale | 87 [43 to 100] | 94 [67 to 100]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03794700/Prot_SAP_000.pdf